CLINICAL TRIAL: NCT06160310
Title: Tuberous Sclerosis Complex and Lymphangioleiomyomatosis Pregnancy Registry
Brief Title: Tuberous Sclerosis Complex and Lymphangioleiomyomatosis Pregnancy Registry (TSC-LAM Registry)
Status: Recruiting | Type: Observational
Sponsor: David M. Ritter (Other)
Responsible Party: Sponsor-Investigator, David M. Ritter, Sponsor/Principal Investigator, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: 2022-0973
Record Dates: First submitted 2023-10-16; First posted 2023-12-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Tuberous Sclerosis Complex; Lymphangioleiomyomatosis
Keywords: Tuberous Sclerosis Complex; TSC; Lymphangioleiomyomatosis; LAM
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational registry designed to gather information about Tuberous Sclerosis Complex (TSC) and Lymphangioleiomyomatosis (LAM) in pregnant women and their child.

DETAILED DESCRIPTION:
Tuberous sclerosis complex (TSC) is caused by mutations in tuberous sclerosis complex 1 (TSC 1) and tuberous sclerosis complex 2 (TSC 2) leading to overactivation of the mammilian target of rapamycin (mTOR) pathway resulting in multiorgan disease. Specifically, patients are at risk for autism, epilepsy, intellectual disability, renal cysts, tuberous sclerosis associated neuropsychiatric disorder (TAND), lymphangioleiomyomatosis (LAM), and benign tumors throughout the body including subependymal giant cell astrocytomas (SEGAs), renal and liver angiomyolipomas (AMLs), and cardiac rhabdomyomas (rhabdomyomas).

Sporadic LAM occurs mostly in women and many patients with LAM have TSC gene mutations.

The purpose of this study is to gather information to help clinicians develop evidence-based guidance for the care of TSC and LAM patients during pregnancy and to provide screening recommendations for fetal TSC.

Participants will be asked to complete monthly online surveys screening for changes in the pregnancy, maternal health/medication changes, and other care. For infants enrolled after birth, clinical data will be collected and reviewed for up to 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A pregnant woman with a clinical or genetic diagnosis of TSC as determined by the 2021 Consensus Guidelines (1)
* A pregnant woman with a diagnosis of LAM
* A pregnant woman with a variant of uncertain significance in TSC 1 or TSC 2
* A pregnant woman who is pregnant and the fetus has a 50% chance of TSC as deemed by the PI or Sub-Is
* A pregnant woman whose fetus is found to have concern for TSC secondary to rhabdomyomas, tubers, or congenital subependymal giant cell astrocytoma.
* An infant born to an enrolled individual.

Exclusion Criteria:

* A pregnant woman without TSC who has used preimplantation genetic testing for TSC unless qualifies under inclusion criteria #4.
* Infants diagnosed with TSC whose birth mother was not enrolled.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This registry is designed to enroll pregnant women who have a TSC and/or LAM diagnosis, a variant of uncertain significance in the TSC 1 or TSC 2 genes, whose fetus has a 50% chance of TSC as deemed by the study PI or Sub-Is, or whose fetus is found to have concern for TSC based on fetal testing.
  Infants born to an enrolled individual regardless of gender and TSC status are eligible for enrollment into the registry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety of mTOR inhibitor in Pregnancy -- mTOR inhibitor adherence | During pregnancy (up to 40 weeks) through 6 months post-delivery
  Assess number of days participant takes mTOR inhibitor in relation to number of days participant was supposed to take mTOR inhibitor.
Safety of mTOR inhibitor in Pregnancy -- mTOR inhibitor dosing | During pregnancy (up to 40 weeks) through 6 months post-delivery
  Review mTOR inhibitor dosing for each participant.
Safety of mTOR inhibitor in Pregnancy -- side effects | During pregnancy (up to 40 weeks) through 6 months post-delivery
  Monitor side effects of mTOR inhibitor experienced by participant.
Maternal-Fetal Complications in TSC | During pregnancy (up to 40 weeks)
  Screening for changes in pregnancy, maternal health/medication changes and other care by using a study-developed monthly questionnaire inquiring about pregnancy status, maternal and/or fetal testing, changes to maternal and fetal care clinical providers, addition or removal of medications, changes in medication doses, and addition of new complications to mother and/or fetus using a list of common gestational complications within prior month.
Maternal Post-Partum Behavioral Health | Post-partum up to 6 months
  Participant will complete Tuberous Sclerosis Complex associated Neuropsychiatric Disorders (TAND) questionnaire.
Maternal Post-Partum Mental Health | Post-partum up to 6 months
  Participant will complete the Edinburgh Postnatal Depression Scale (EPDS).
Optimum Time of Fetal Imaging for TSC | Birth through 5 years of Age
  Compare fetal imaging to imaging and clinical data including echocardiograms, electrocardiograms, genetic testing results, magnetic resonance images of the brain and abdomen, ultrasounds.

CONTACTS AND LOCATIONS:
Overall Officials: David M Ritter, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States